CLINICAL TRIAL: NCT02011425
Title: The Effects of Mandibular Advancement Appliance Therapy on Masseter Muscle Activity During Sleep in Obstructive Sleep Apnea Patients: a Study in Clinical Practice
Brief Title: The Effects of Oral Appliance Therapy on Masseter Muscle Activity in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Nelly Huynh, Professor, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 13-105-CERES-D; NH-13-SP-MassActivity (Other: Faculte de medecine dentaire, Universite de Montreal)
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; oral appliance; therapy; masseter muscle activity; randomized controlled trial; mandibular advancement device; mandibular advancement appliance; arousals
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mandibular advancement appliance (Experimental): mandibular advancement appliance (SomnoDent by SomnoMed)
  Interventions: Device: mandibular advancement appliance
- without mandibular advancement appliance (No Intervention): no therapy

INTERVENTIONS:
Device: mandibular advancement appliance — mandibular advancement appliance
  Other Names: mandibular advancement splint; oral appliance; mandibular repositioning splint; mandibular repositioning appliance
  Arms: mandibular advancement appliance

SUMMARY:
Previous studies have shown that contractions of the jaw-closing masseter muscle (MAS) often occur shortly after respiratory events during sleep in obstructive sleep apnea (OSA) patients. Although it has been hypothesized that such non-specific motor activations may contribute to restoration of a compromised upper airway during respiratory events, proper physiological understanding of MAS contractions in patients with OSA is lacking. MAS contractions are usually associated with the termination of respiratory events, but these contractions do not always occur after respiratory events. Therefore, the above-stated hypothesis that "non-specific motor activations of the jaw-closing masseter muscle (MAS) may contribute to restoration of a compromised upper airway during respiratory events" is not accepted yet. Further, Kato et al. concluded from a recent study that MAS contraction is an orofacial manifestation of a general motor reaction to arousal occurring during sleep in OSA patients. This suggests that MAS contraction after a respiratory event is dependent on the arousal response rather than on the respiratory events per se.

DETAILED DESCRIPTION:
OSA patients will be invited for participation in this study when they fulfil the predetermined inclusion criteria and exclusion criteria. The number of OSA patients that will be included for this study will be 25 based on a power analysis with a power of 80% and a significance level of 5% (two-sided). Informed consent will be obtained by signing form approved by the ethics board of the Université de Montréal.

The patients will be instructed to wear the mandibular advancement appliance (MAA) every night upon delivery. After a habituation period of three to six months patients will undergo two follow-up polysomnographic (PSG) recordings (see below).

The study has a randomized controlled crossover design, in which two experimental conditions (with MAA in situ versus without MAA in situ) will be compared in random order. A washout period of one week will be used for the MAA therapy.The study consists of three PSG recordings per patient: a baseline recording for the inclusion/exclusion of patients, and two follow-up recordings. The first and second follow-up nights will be used to establish, in a random order, the baseline for masseter muscle activity and arousals, and the effects of the MAA on these parameters. The two follow-up recordings will be performed within one week.

The ambulatory follow-up PSG recordings will be obtained at home. The mounting will be performed by a trained sleep technician. PSG recordings are made using surface electrodes according to the standard technical protocol used in previous OSA studies at the same laboratory.

The PSG recordings will be scored manually in 30-s epochs, and standard sleep and respiratory outcome variables will be obtained. All data analyses will be performed under blind conditions for the PSG recordings (with or without an MAA in situ) by one technician.

ELIGIBILITY:
Inclusion Criteria:

* age between 30-65 years
* OSA patients with an apnea-hypopnea index (AHI) between 15 and 45 events per hour, and a report of excessive daytime sleepiness (Epworth Sleepiness Score > 10) or at least two of the symptoms suggested by the American Academy of Sleep Medicine Task Force, e.g., unrefreshing sleep and daytime fatigue.

Exclusion Criteria:

* Evidence of respiratory/sleep disorders other than OSA
* a Body Mass Index (BMI) > 40, medication usage that could influence respiration or sleep
* reversible morphological upper airway abnormalities (e.g., enlarged tonsils)
* severe temporomandibular disorders
* untreated periodontal problems or dental pain
* a lack of retention possibilities for an MAA

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
number of masseter muscle activity events | up to 6 month following start of use of mandibular advancement appliance
  Motor activations in the masseter muscle during sleep will be scored when the EMG level is at least 10% of the maximum voluntary contraction (MVC) established before sleep.

SECONDARY OUTCOMES:
rhythmic masticatory muscle activity index | up to 6 month following start of use of mandibular advancement appliance
  Number of rhythmic masticatory muscle activity per hour of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Huynh, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li D, Aarab G, Lobbezoo F, Arcache P, Lavigne GJ, Huynh N. The effects of mandibular advancement appliance therapy on the sequence of jaw-closing muscle activity and respiratory events in individuals with obstructive sleep apnea. Sleep Breath. 2023 May;27(2):757-764. doi: 10.1007/s11325-022-02624-z. Epub 2022 Apr 28. PMID 35484327
- [Derived] Li D, Aarab G, Lobbezoo F, Arcache P, Lavigne GJ, Huynh N. Accuracy of sleep bruxism scoring based on electromyography traces of different jaw muscles in individuals with obstructive sleep apnea. J Clin Sleep Med. 2022 Jun 1;18(6):1609-1615. doi: 10.5664/jcsm.9940. PMID 35212262
- [Derived] Aarab G, Arcache P, Lavigne GJ, Lobbezoo F, Huynh N. The effects of mandibular advancement appliance therapy on jaw-closing muscle activity during sleep in patients with obstructive sleep apnea: a 3-6 months follow-up. J Clin Sleep Med. 2020 Sep 15;16(9):1545-1553. doi: 10.5664/jcsm.8612. PMID 32501212